CLINICAL TRIAL: NCT03210922
Title: Effect of Semirigid Cervical Collar During Nasotracheal Intubation by Glidescope in the Elective Cervical Spinal Surgical Patients: a Study of Clinical Predictors and Outcomes
Brief Title: Semirigid Cervical Collar and Nasotracheal Intubation by Glidescope in Cervical Spine Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, vghtpe user, Principal Investigator, Associate Professor, Taipei Veterans General Hospital, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2017-06-009B
Record Dates: First submitted 2017-06-19; First posted 2017-07-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Orthosis
Keywords: cervical collar, nasoendotracheal intubation, glidescope

STUDY DESIGN:
Intervention Model Description: The patients are randomized into one of the two group: the collar group or the non-collar group before anesthetic induction. In the collar group, the patient was put on a Miami cervical collar and then anesthetic induction and nasotracheal intubation are performed. the non-collar group receive the same anesthetic care without a collar as a control.
Who Masked: Outcomes Assessor
Masking Description: The anesthetic induction and nasotracheal induction are performed by one anesthesiologist. Another anesthesiology calculated the intubation time according to the video recording.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Collar group (Experimental): Standard of anesthetic care and nasointubation with patient wearing the Miami cervical collar.
  Interventions: Device: Miami cervical collar
- Non-collar group (No Intervention): Standard of anesthetic care and nasointubation with patient not wearing the Miami cervical collar.

INTERVENTIONS:
Device: Miami cervical collar — Collar group is put on the Miami cervical collar.
  Arms: Collar group

SUMMARY:
Effect of semirigid cervical collar during nasotracheal intubation by Glidescope in the elective cervical spinal surgical patients: a study of clinical predictors and outcomes

DETAILED DESCRIPTION:
Clinically used cervical orthoses can effectively limit cervical spine motion in all direction and provide protection. Among them, the restriction by Miami semirigid collar was superior, with the least tissue-interface pressure of neck. It is one of the most used semirigid collars for patients' protection in the operating theatre. However, the presence of the semirigid collar was shown to result in a poorer view at laryngoscopy, possibly due to a reduction in mouth opening. Nasotracheal intubation is sometimes applied in cervical spinal surgeries for those receiving anterior approach for a higher cervical spine (C3) level, and/ or combined with a short neck, or due to surgeon's preference. Glidescope minimizes cervical movements during laryngoscopy, facilitates nasotracheal intubation than direct laryngoscopy and requires less technical skill than fiberoptic tracheal intubation. The investigation was to assess the effect of cervical collar on nasotracheal intubation and potential hazard factors of prolonged time for nasotracheal intubation with Gildescope in patients scheduled for elective cervical spinal surgery.

ELIGIBILITY:
Inclusion Criteria:

* elective cervical spine surgery
* scheduled for nasotracheal intubation
* not requiring orthosis for prophylactic protection

Exclusion Criteria:

* Risk of pulmonary aspiration of gastric contents
* Pathology of the nasal cavity
* Abnormal coagulation function
* Extensive and severe cord compression
* Refused to sign informed consent.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2017-07-13 (Actual); Primary Completion 2018-04-13 (Actual); Study Completion 2018-04-18 (Actual)

PRIMARY OUTCOMES:
Nasointubation Time | Intraoperative
  intubation time assisted by Glidescope

SECONDARY OUTCOMES:
subjective scoring of ease of intubation | Intraoperative
  ease of intubation scored with visual analogue scale
magill forceps for nasointubation | Intraoperative
  whether magill forcepts is required to facilitate nasointubation

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Cheng Huang, M.D., Ph.D., Principal Investigator — Center of Neural Regeneration, Department of Neurosurgery, Neurological Institute, Taipei Veterans General Hospital
Locations (1):
- Taipei Veterans General Hospital, Taipei, Beitou, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided